CLINICAL TRIAL: NCT04802265
Title: To Compare Anatomical and Functionnal Outcomes in Patients Undergoing Epiretinal Membrane Surgery With and Without Internal Limiting Membrane Peeling
Brief Title: EpiRetinal Membrane Peeling and Internal Limiting Membrane
Acronym: ERMP&ILM
Status: Terminated | Type: Observational
Why Stopped: departure of the intern in charge of the study
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RBHP 2021 SILLAIRE; 2021-A00071-40 (Other: 2021-A00071-40)
Record Dates: First submitted 2021-03-10; First posted 2021-03-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Epiretinal Membrane; Macular Pucker; Internal Limiting Membrane
Keywords: Epiretinal membrane; Epiretinal membrane peeling; Macular pucker; Internal limiting membrane (ILM) peeling; Pars plana vitrectomy
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ILM peeling: ILM is peeled during epiretinal membrane surgery
  Interventions: Procedure: Epiretinal membrane surgery
- without ILM peeling: ILM is not peeled during epiretinal membrane surgery
  Interventions: Procedure: Epiretinal membrane surgery

INTERVENTIONS:
Procedure: Epiretinal membrane surgery — The surgery consists of a 23 or 25-gauge pars plana vitrectomy (PPV). The surgery was performed peri-bulbar anesthesia and could be combined with phacoemulsification.
  An intraocular dye is used to well visualized and facilitate ERM peeling. The ILM is not actively peeled. A search for iatrogenic breaks is performed towards the end of the procedure. Areas suspicious for breaks are treated with cryotherapy or peripheral endolaser.

SUMMARY:
To study and compare visual acuity in patients undergoing removal of the epiretinal membrane with and without the removal of the internal limiting membrane at baseline versus 6 month.

DETAILED DESCRIPTION:
This prospective cohort study includes 2 arms : with and without internal limiting membrane (ILM) peeling.

Each patient undergo the same procedure : first of all pars plana vitrectomy, then internal limiting membrane peeling is performed and facilitated by the use of dye, which aids in better visualization of the ILM.

If the ILM is removed in same time : the patient is ranked in the "ILM peeling" group If the ILM is not removed : the patient is ranked in the "non ILM peeling" group.

If the ILM is partially removed, the patient is not enrolled.

The outcomes are recorded for 6 months : at baseline, day 15, 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* adult up to 18 years old,
* diagnosed and treated surgically

Exclusion Criteria:

* proliferative diabetic retinopathy,
* ocular trauma,
* central veinous occlusion,
* intra-ocular tumor, total retinal detachment,
* central visual field loss in glaucomatous patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult diagnosed for epiretinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) (metric : LogMAR) | prior to surgery
  BCVA is measured at each medical appointment. Monoyer Scale is used and results are converted in LogMAR scale.
Best corrected visual acuity (BCVA) (metric : LogMAR) | Day 180
  BCVA is measured at each medical appointment. Monoyer Scale is used and results are converted in LogMAR scale.

SECONDARY OUTCOMES:
BCVA at day 15, 1, 3 month. | Day 15, Day 30, Day 90
  BCVA is measured at each medical appointment. Monoyer Scale is used and. Resulats are converted in LogMAR scale.
near visual acuity measured at baseline, day 15, 1, 3 and 6 month | Day 180
  near visual acuity is measured at each medical appointment using Parinaud Scale
central retinal thickness (CRT) | Day 180
  CRT is measured on optical coherence tomography (OCT) at baseline, day 15, 1 , 3 and 6 months
peeling initiation retinal thickness | Day 180
  to evaluate the damage due to the membrane gripping during the peeling initiation, retinal thickness is performed at this location by OCT.
10° visual field | Day 180
  a 10° Visual Field is performed at baseline, 1 month and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Sillaire, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, AURA, France